CLINICAL TRIAL: NCT04082325
Title: Interventional, Randomized, Double-blind, Sequential-group, Placebo-controlled, Single-ascending-oral-dose Study Investigating the Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Properties of Lu AF88434 and Open-label Crossover Study to Investigate the Intra-individual Variability, Metabolic Profile, and Effect of Food on Lu AF88434 in Healthy Young Men
Brief Title: Study Investigating the Safety and Tolerability of Lu AF88434 in Healthy Young Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 18144A
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A Lu AF88434 or Placebo (Experimental): 6 cohorts (cohort A1 to A6) with 9 subjects in each cohort. In each cohort 6 subjects will receive single doses of Lu AF88434 and 3 subjects will receive placebo
  Interventions: Drug: Lu AF88434; Drug: Placebo
- Part B1 Lu AF88434 Fed-Fasting-Fasting (Experimental): 4 subjects will receive an identical oral dose of Lu AF88434 in Group B1. The treatment sequence for Group B1 is: Fed-Fasting-Fasting. 14C-spiked dose (Lu AF99723) will be given in the last treatment sequence.
  Interventions: Drug: Lu AF88434; Drug: Lu AF99723 14C spiked dosage ([14C]-radiolabelled Lu AF88434)
- Part B2 Lu AF88434 Fasting-Fed-Fasting (Experimental): 4 subjects will receive an identical oral dose of Lu AF88434 in Group B2. The treatment sequence for Group B2 is: Fasting-Fed-Fasting. 14C-spiked dose (Lu AF99722) will be given in the last treatment sequence.
  Interventions: Drug: Lu AF88434; Drug: Lu AF99722 14C spiked dosage ([14C]-radiolabelled Lu AF88434)
- Part B3 Lu AF88434 Fasting-Fasting-Fed (Experimental): 4 subjects will receive an identical oral dose of Lu AF88434 in Group B3. The treatment sequence for Group B3 is: Fasting-Fasting-Fed.
  Interventions: Drug: Lu AF88434

INTERVENTIONS:
Drug: Lu AF88434 — Lu AF88434, single oral solution Starting dose will be 0.2 mg, actual doses for following cohorts will be defined based on results from preceding dosing group(s).
Drug: Lu AF99722 14C spiked dosage ([14C]-radiolabelled Lu AF88434) — Oral solution
  Arms: Part B2 Lu AF88434 Fasting-Fed-Fasting
Drug: Lu AF99723 14C spiked dosage ([14C]-radiolabelled Lu AF88434) — Oral solution
  Arms: Part B1 Lu AF88434 Fed-Fasting-Fasting
Drug: Placebo — Placebo to Lu AF88434 oral solution, single dose
  Arms: Part A Lu AF88434 or Placebo

SUMMARY:
This study evaluates the effect of Lu AF88434 on the body and what the body does to Lu AF88434 and the effect of food after swallowing single oral doses

ELIGIBILITY:
Inclusion Criteria:

-Healthy young non-smoking men with a body mass index (BMI) ≥18.5kg/m2 and ≤30kg/m2 at the Screening Visit and Baseline Visit.

Exclusion Criteria:

* The subject has or has had any clinically significant immunological, cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, or psychiatric disease or other major disorder.
* For Part B: The subject has received radiolabelled material <12 months prior to the Screening Visit.

Other inclusion and exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events | From screening to Day 11
  Safety and tolerability based on the safety assessments (clinical safety laboratory tests, vital signs, weight, ECG parameters)
Cmax Lu AF88434 | From 0 to 96 hours
  Maximum observed plasma concentration
AUC(0-inf) Lu AF88434 | From 0 to 96 hours
  Area under the plasma concentration time curve from zero to infinity
CL/F Lu AF88434 | From day 1 to day 5
  Oral clearance for Lu AF88434 in plasma
Cumulative recovery of radioactivity in urine, faeces, and total (urine+faeces) (% of administered dose) | From 0 to Day 14
Total recovery of radioactivity in urine, faeces, and total (urine+faeces) (% of administered dose) | From 0 to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- QPS, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided